CLINICAL TRIAL: NCT07193732
Title: The Application of Islamically Integrated Chair-Work Techniques For Unfinished Business in Patients With Prolonged Grief
Brief Title: Islamically Integrated Chair-Work for Bereaved Muslims
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E-71395021-050.06.04-35013
Record Dates: First submitted 2024-03-06; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Grief; Emotion Regulation; Bereavement
Keywords: loss; bereavement; grief; unfinished bussines
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2-weeks baseline (Experimental): Participants will wait for a two-week period before starting psychotherapy sessions, during which time they will complete questionnaires. Following this period, they will engage in a 7-week psychotherapy process.
  Interventions: Behavioral: Psychotherapy-Empathic Attunement Phase; Behavioral: Psychotherapy - Chair-work intervention phase; Behavioral: Psychotherapy - Cognitive consolidation and spiritually behavioral activation phase
- 4-weeks baseline (Experimental): Participants will wait for a four-weeks period before starting psychotherapy sessions, during which time they will complete questionnaires. Following this period, they will engage in a 7-week psychotherapy process.
  Interventions: Behavioral: Psychotherapy-Empathic Attunement Phase; Behavioral: Psychotherapy - Chair-work intervention phase; Behavioral: Psychotherapy - Cognitive consolidation and spiritually behavioral activation phase
- 6-weeks baseline (Experimental): Participants will wait for a six-week period before starting psychotherapy sessions, during which time they will complete questionnaires. Following this period, they will engage in a 7-week psychotherapy process.
  Interventions: Behavioral: Psychotherapy-Empathic Attunement Phase; Behavioral: Psychotherapy - Chair-work intervention phase; Behavioral: Psychotherapy - Cognitive consolidation and spiritually behavioral activation phase

INTERVENTIONS:
Behavioral: Psychotherapy-Empathic Attunement Phase — The initial focus of our therapeutic intervention is on establishing empathic attunement to aid individuals in processing the inherent pain of grief in a constructive manner. For this phase, therapists will focus solely on adhering to the relationship formation and introspective exploration. Practitioners aimed at empathetically tuning into the patient's emotional experience, validating and reassuring the patient's emotional state, and adhering to the fundamental principles of empathy, sincerity, and positive regard for establishing and upholding a strong therapeutic alliance. Also, accompanying the patients to uncover and process the natural pain to gain self-awareness about their emotions.
Behavioral: Psychotherapy - Chair-work intervention phase — During this phase, bereavement person will conduct imaginal conversation with a deceased. Practitioners utilized the resolution model including 5 components: (1) emotional reaction of the bereavement (blame, hurt, regret etc.) and enactment of the deceased; (2) differentiation of the bereavement's feelings and deceased's specific negative aspects accessed; (3) intense expression of the bereavement's specific emotions; (4) expression of the bereavement's previously unmet interpersonal needs from the deceased and the deceased validates bereavement's feelings; (5) understanding and forgiveness of the deceased or shift in view of the deceased.
Behavioral: Psychotherapy - Cognitive consolidation and spiritually behavioral activation phase — Cognitive consolidation and spiritually behavioral activation complement the emotional interventions implemented in earlier stages. This cognitive process aids in the transformation and integration of adaptive growth, enabling patients to assimilate the knowledge and insights acquired during therapy. Therapists take a directive and co-constructivist approach, guiding patients to discover emotionally adaptive reconciliations and meanings that challenge and reshape their emotional and cognitive frameworks in the cognitive consolidation and spiritually behavioral activation phase. Aligned with this cognitive shift, spiritual behavioral activations involve creating plans to address unmet needs.

SUMMARY:
This study aims to develop and to evaluate the efficacy of an Islamically integrated chair-work intervention designed to assist Muslims experiencing prolonged grief in resolving unfinished business tension. Employing a randomized, non-concurrent, multiple baseline design, the study comprises five phases: (1) baseline assessment, (2) empathic attunement, (3) Traditional Islamically Integrated Psychotherapy (TIIP) chair-work intervention, (4) cognitive consolidation & spiritually behavioral activation, and (5) follow-up. By integrating insights from early Islamic scholars like Al-Kindi, Abu Bekir er-Razi, and Ibn Sina, alongside psychological counseling and cultural elements, this intervention aims to fill a crucial gap in existing literature. Grief, a normal emotional reaction after the loss of a loved one, is typically resolved over time without professional intervention. However, a small yet significant number of individuals experience prolonged grief disorder (PGD), a persistent and impairing form of grief lasting over 6 months. Unfinished business, indicating unresolved relational issues with the deceased, is a key risk factor for severe PGD. Higher levels of unfinished business are associated with increased psychological problems and unhealthy expressions of grief. Within the framework of Traditional Islamically Integrated Psychotherapy (TIIP), unfinished business is viewed as an emotionally charged problem. Processing this emotional burden during TIIP sessions aims to facilitate resolution, replacing maladaptive emotions with adaptive ones, fulfilling emotional needs, and establishing new meanings for unresolved conflicts. Sense-making of one's loss is crucial for a healthier grieving process, making meaning-oriented techniques more effective in grief therapy. Moreover, research indicates that the expression of grief is influenced by spirituality, religious beliefs, and practices. Yet, there is a lack of faith-based intervention programs tailored for grieving Muslims. This study seeks to address this gap by providing closure and therapeutic methods that cater to the nuanced emotional struggles of bereaved Muslims, offering a faith-based approach previously unavailable in the literature.

DETAILED DESCRIPTION:
This study explores the effectiveness of the Islamically Integrated chair-work techniques for unfinished business in patients with prolonged grief. Grief is characterized by intense emotional suffering, a yearning or longing for the deceased, a sense of shock or shock at the loss, and difficulty in moving on after the loss. The loss of a loved one is an unavoidable, universal life experience, although it is also one of the most stressful. Mourning individuals often become accustomed to the death of a loved one over time, but a small yet significant number of people subsequently experience serious psychological problems. Individuals who have experienced the loss of a loved one have a higher risk of developing psychopathology in the first year after bereavement, including an increased risk of self-harm and a higher risk of suicide. This group is also susceptible to a high degree of morbidity and mortality.

Studies over the last few decades suggest that many grieving individuals experience persistent difficulties associated with bereavement that exceeds the expected social, cultural, or religious expectations. With the publication of the DSM-5-TR (The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision), the term Prolonged Grief Disorder (PGD) has been coined for those experiencing grief after the loss of a loved one, lasting longer than 12 months for adults or 6 months for children, and causes significant impairment. An estimated 7%-10% of bereaved adults will experience the persistent symptoms of prolonged grief disorder. Among children and adolescents who have lost a loved one, approximately 5%-10% will experience depression, posttraumatic stress disorder (PTSD), and/or prolonged grief disorder following the bereavement. Although only a minority of grievers suffer from some psychological problems, misdiagnoses have been common because there was no specific diagnosis for grief in the past.

One of the most important risk factors for severe PGD is unfinished business, which indicates incomplete, unexpressed, or unresolved relational issues with the deceased. It was found that 43% of bereaved individuals exhibit some degree of unfinished business. Higher levels of unfinished business are associated with higher levels of psychological problems and unhealthy ways of expressing grief. In the context of the Traditional Islamically Integrated Psychotherapy (TIIP) framework, unfinished business is conceptualized as an emotionally-charged problem. Through the emotional processing of unfinished business during TIIP psychotherapy sessions, suffering patients are able to find a resolution to their emotional problems, which leads to the replacement of maladaptive emotions with more adaptive ones, need fulfillment, and the creation of new meanings for unresolved conflicts. Indeed, making sense of one's loss is associated with a healthier grieving process. Therefore, meaning-oriented techniques are more effective in grief therapy. Furthermore, the results of a systematic literature review show that the expression of grief is directly influenced by spirituality, religious beliefs, and practices. Yet, there is no intervention program specifically designed for grieving Muslims that is faith-based. From an Islamic perspective, death is seen as a natural part of the human lifecycle, including the soul's transfer from this world to the after-world.

In order to better explain the mourning process, a number of theories have been put forth in Western literature. Nevertheless, they largely ignore socio-cultural variations outside of the bereavement of white people in Europe or North America. Although it is known that religion and belief have a very important role in the mourning experience, there are no intervention programs specifically tailored for grieving Muslims that utilize a faith-based approach reported in the literature. This study aims to develop and explore the utility of an Islamically integrated chair-work intervention to help resolve unfinished business for Muslims who have experienced prolonged grief. A randomized, non-concurrent, multiple baseline design is planned for the proposed study to use Islamically integrated chair-work intervention using five phases: (1) baseline phase, (2) empathic attunement phase, (3) TIIP -Traditional Islamically Integrated Psychotherapy- chair-work intervention phase, (4) cognitive consolidation & spiritually behavioral activation phase, and (5) follow-up phase (1 month post). The protocol will be implemented on a weekly basis through 50-minute, face-to-face individual psychotherapy sessions, totaling seven sessions.

In this study, the multiple-baseline design comprises five phases, with the initial phase designated as the baseline. Notably, the duration of this baseline phase will be randomly varied among participants. This random allocation to baseline periods of different lengths facilitates the evaluation of whether symptom changes are specifically associated with the application of the intervention. Participants will be randomly assigned to one of three baseline lengths-2, 4, or 6 weeks-allowing for varied observation periods before the intervention commences. During the baseline phase, participants will complete the primary outcome measurement. This study will demonstrate the utilization of the Islamically integrated chair-work in assisting bereaved Muslims facing numerous psychological, physiological, social, and economic risks to resolve the unfinished business on account of their prolonged grief. The Islamic integration of the chair-work intervention incorporates insights from early Islamic thinkers with psychological counseling and cultural and religious elements.

Early Islamic scholars such as Al-Kindi, Abu Bekir al-Razi, and Ibn Sina had conceptualized grief and sorrow and provided strategies to cope with the emotional struggles following the loss of a loved one. The investigators have integrated certain therapeutic methods from early Islamic scholars to address the challenges of grief after a loss. Al-Kindi begins by defining sorrow and offering guidance for those suffering from grief. His definition emphasizes sorrow arising from losing a loved object, conceptualized as "loss," and also from unfulfilled desires, conceptualized as "missing out." Al-Kindi's concept of "loss" resonates with the empathic attunement process in the Islamically integrated psychotherapy protocol. The 'missing out' forms the basic framework of unfinished business after loss. The investigators integrated the concept of "grief meditation" chair-work intervention to resolve unfinished business tension from al-Razi's advice to imagine the scenarios of loss. Finally, a phase of cognitive consolidation and spiritually behavioral activation draws influence from Ibn Sina's teachings. He posited that due to the obscurity of death, individuals struggle to establish a healthy relationship with the concept of death. For the final part of the protocol, patients search for meaning from the loss with the therapist, then transform cognitive and emotional schemas and devise behavioral plans based on newly acquired perspectives and emotions. The importance of the study stems from an Islamically integrated interventional method of providing closure to individuals experiencing prolonged grief that is otherwise not available in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Loss of a loved one 6 months to 5 years ago,
* Grieving for unresolved tension for a loved one (24 or more points on the Unfinished Business in Bereavement Scale),
* Religiously adherent adults (according to self report)

Exclusion Criteria:

* Imminent suicide risk or self-harm,
* Current substance or alcohol dependence,
* Past or current psychotic disorders or bipolar disorder;
* Currently receiving any form of psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The Unfinished Business in Bereavement Scale - Brief | Baseline, weekly through Week 7 (end of treatment), and at 1-month follow-up (up to 11 weeks total)
  The Unfinished Business in Bereavement Scale - Brief (UBBS - Brief) is a self-report measurement tool developed by Holland et al. (2020). Utilizing a 5-point Likert scale (ranging from 1 = Not at all distressed to 5 = Extremely distressed), the UBBS - Brief comprises 8 items and includes two subscales: 'unfulfilled wishes' and 'unresolved conflict.'
Prolonged Grief Disorder-13 Scale | Baseline (Week 0), end of treatment (Week 7), and 1-month follow-up (Week 11; up to 11 weeks total).
  The Prolonged Grief Disorder-13 (PG-13) Scale, developed by Prigerson et al. (2009) serves as a diagnostic tool for prolonged grief disorder (PGD) and aims to assess the severity of symptoms experienced after a loss. PG-13 comprises a total 13 item, with 11 of them utilizing 5-Likert point scale (1 = Not at all, 3= At least once a week, 5= Several times a day) to gauge severity of the struggles associated with the loss. And the remaining two items are yes/no question to designed to determine the duration time post-loss (a minimum of 6 months) and to assess dysfunction criterion. An increase in the cumulative scores obtained from the 11 items on the scale indicates a rise in the severity of prolonged grief symptoms. The PG-13 outlines five criteria (A-E) to diagnose PGD: (A) event criterion; (B) separation distress; (C) Duration Criterion; (D) cognitive, emotional, and behavioral symptoms; and (E) impairment criterion (Prigerson et al., 2009).
The Grief Cognitions Questionnaire | Baseline (Week 0), end of treatment (Week 7), and 1-month follow-up (Week 11; up to 11 weeks total).
  The Grief Cognitions Questionnaire (GCQ) was developed by Boelen et al. (2003) comprises a 38-item self-report assessment tool utilizing a 6-point Likert scale (ranging from 0 = strongly disagree to 5 = strongly agree) encompassing nine distinct subscales. Its primary function is to evaluate the negative cognitions experienced by bereaved individuals following a loss, which may contribute to the complexity of the grieving process. The Turkish version includes 30 items, consolidating into six subscales (Cesur and Durak-Batıgün, 2018): (1) negative cognitions about future after loss, (2) negative/threatening interpretation of emotions and reactions to loss, (3) negative cognitions about self after loss, (4) negative cognitions about world after loss, (5) cherish grief and, (6) negative cognitions about others after loss. Scores on the questionnaire range from 0 to 150, with higher scores indicating a greater intensity of negative cognitions.

SECONDARY OUTCOMES:
The Client Emotional Arousal Scale III | Baseline (Week 0), end of treatment (Week 7), and 1-month follow-up (Week 11; up to 11 weeks total).
  The Client Emotional Arousal Scale III (CEAS-III), devised by Warwar and Greenberg in 1999, is an observer-rated measure designed to assess the depth and intensity of clients' emotional expressions. This scale examines emotional arousal by analyzing both vocal and bodily cues, utilizing a 7-point scale to rate the intensity of expressed emotions. CEAS-III focuses on primary emotions, including anger, fear, joy, love, sadness, and surprise, and differentiates emotional levels, ranging from lower levels (1-3) indicating limited emotional arousal to higher levels (4-7) representing increased intensity. Level 4 signifies moderate arousal with noticeable disruptions in speech patterns due to emotional overflow, while level 7 indicates an extremely intense and uncontrollable emotional state, resulting in a significant disruption of usual speech patterns.
Patient Health Questionnaire-9 | Baseline (Week 0), end of treatment (Week 7), and 1-month follow-up (Week 11; up to 11 weeks total).
  The Patient Health Questionnaire - 9 (PHQ-9) was developed by Kroenke et al. (2001) to diagnose depression and measure severity of depression and comprises nine items, self-report assessment tool utilizing a four-point Likert scale (ranging from 0 = not at all, to 3 = nearly every day). Scores on the questionnaire range from 0 to 27, with a cut-off point of 10, higher scores indicating a severity of depressive symptoms
Generalized Anxiety Disorder-7 | Baseline (Week 0), end of treatment (Week 7), and 1-month follow-up (Week 11; up to 11 weeks total).
  The Generalized Anxiety Disorder - 7 (GAD-7) was developed by Spitzer et al. (2006) to diagnose generalized anxiety and measure severity of generalized anxiety and comprises seven items, self-report assessment tool utilizing a four-point Likert scale (ranging from 0 = not at all, to 3 = nearly every day). Scores on the questionnaire range from 0 to 21, higher scores indicating a more severe generalized anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Keshavarzi, Psy.D., Study Chair — Ibn Haldun University
Locations (1):
- Ibn Haldun University, Istanbul, Başakşehir, Turkey (Türkiye)

REFERENCES:
- [Background] Prigerson HG, Horowitz MJ, Jacobs SC, Parkes CM, Aslan M, Goodkin K, Raphael B, Marwit SJ, Wortman C, Neimeyer RA, Bonanno GA, Block SD, Kissane D, Boelen P, Maercker A, Litz BT, Johnson JG, First MB, Maciejewski PK. Prolonged grief disorder: Psychometric validation of criteria proposed for DSM-V and ICD-11. PLoS Med. 2009 Aug;6(8):e1000121. doi: 10.1371/journal.pmed.1000121. Epub 2009 Aug 4. PMID 19652695
- [Background] Holland JM, Klingspon KL, Lichtenthal WG, Neimeyer RA. The Unfinished Business in Bereavement Scale (UBBS): Development and psychometric evaluation. Death Stud. 2020;44(2):65-77. doi: 10.1080/07481187.2018.1521101. Epub 2018 Dec 4. PMID 30513256
- [Background] Boelen, P. A., & Lensvelt-Mulders, G. J. Psychometric properties of the grief cognitions questionnaire (GCQ). Journal of Psychopathology and Behavioral Assessment. 2005; 27(4): 291-303.
- [Background] Warwar, S., & Greenberg, L. S. Client emotional arousal scale-III. Unpublished manuscript, York University, Toronto, Ontario, Canada. 1999
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Papa A, Lancaster NG, Kahler J. Commonalities in grief responding across bereavement and non-bereavement losses. J Affect Disord. 2014 Jun;161:136-43. doi: 10.1016/j.jad.2014.03.018. Epub 2014 Mar 25. PMID 24751321
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] Prigerson HG, Boelen PA, Xu J, Smith KV, Maciejewski PK. Validation of the new DSM-5-TR criteria for prolonged grief disorder and the PG-13-Revised (PG-13-R) scale. World Psychiatry. 2021 Feb;20(1):96-106. doi: 10.1002/wps.20823. PMID 33432758
- [Background] Chen Z, Ying J, Ingles J, Zhang D, Rajbhandari-Thapa J, Wang R, Emerson KG, Feng Z. Gender differential impact of bereavement on health outcomes: evidence from the China Health and Retirement Longitudinal Study, 2011-2015. BMC Psychiatry. 2020 Oct 22;20(1):514. doi: 10.1186/s12888-020-02916-2. PMID 33092555
- [Background] Szuhany KL, Young A, Mauro C, Garcia de la Garza A, Spandorfer J, Lubin R, Skritskaya NA, Hoeppner SS, Li M, Pace-Schott E, Zisook S, Reynolds CF, Shear MK, Simon NM. Impact of sleep on complicated grief severity and outcomes. Depress Anxiety. 2020 Jan;37(1):73-80. doi: 10.1002/da.22929. PMID 31916662
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders (5th Ed., Text Rev.).; 2022.
- [Background] Pos AE, Paolone DA, Smith CE, Warwar SH. How does client expressed emotional arousal relate to outcome in experiential therapy for depression? Pers Exp Psychother. 2017;16(2):173-190. doi:10.1080/14779757.2017.1323666
- [Background] Boelen PA, van den Hout MA, van den Bout J. A cognitive-behavioral conceptualization of complicated grief. Clin Psychol Sci Pract. 2006;13(2):109-128. doi:10.1111/j.1468-2850.2006.00013.x
- [Background] Cesur-Soysal G, Durak-Batigun A. Prolonged grief, emotion regulation and loss-related factors: An investigation based on cognitive and behavioral conceptualization. Death Stud. 2022;46(6):1316-1328. doi: 10.1080/07481187.2020.1846639. Epub 2020 Nov 12. PMID 33180665
- [Background] Holland JM, Thompson KL, Rozalski V, Lichtenthal WG. Bereavement-related regret trajectories among widowed older adults. J Gerontol B Psychol Sci Soc Sci. 2014 Jan;69(1):40-7. doi: 10.1093/geronb/gbt050. Epub 2013 Jun 13. PMID 23766434
- [Background] Klingspon KL, Holland JM, Neimeyer RA, Lichtenthal WG. Unfinished Business in Bereavement. Death Stud. 2015;39(7):387-98. doi: 10.1080/07481187.2015.1029143. PMID 26057117
- [Background] Keshavarzi H, Keshavarzi S. Emotionally Oriented Psychotherapy. In: Keshavarzi H, Khan F, Ali B, Awaad R, eds. Applying Islamic Principles to Clinical Mental Health Care. Routledge; 2020:171-208. doi:10.4324/9781003043331-12
- [Background] Holland JM, Neimeyer RA. An examination of stage theory of grief among individuals bereaved by natural and violent causes: a meaning-oriented contribution. Omega (Westport). 2010;61(2):103-20. doi: 10.2190/OM.61.2.b. PMID 20712139
- [Background] De Stefano R, Muscatello MRA, Bruno A, Cedro C, Mento C, Zoccali RA, Pandolfo G. Complicated grief: A systematic review of the last 20 years. Int J Soc Psychiatry. 2021 Aug;67(5):492-499. doi: 10.1177/0020764020960202. Epub 2020 Sep 24. PMID 32972293
- [Background] Beckett C, Dykeman C. A Metatheory of Grief: implications for Counselors. Ideas Res You Can Use. 2017;(30):1-15.
- [Background] Jayyusi-lehn G. The Epistle of Ya'qub ibn Ishaq al-Kindi on the Device for Dispelling Sarrow. 2002;29:121-135. doi:10.1080/135301902200001263
- [Background] Melhem NM, Porta G, Walker Payne M, Brent DA. Identifying prolonged grief reactions in children: dimensional and diagnostic approaches. J Am Acad Child Adolesc Psychiatry. 2013 Jun;52(6):599-607.e7. doi: 10.1016/j.jaac.2013.02.015. Epub 2013 Apr 24. PMID 23702449
- [Background] Ibn Sina, Alî b. Sînâ, Tura, H. Ölüm korkusundan kurtuluş risalesi; Namaz risalesi. orhan Mete ve Ortağı Kollektif Şirketi Matbaası. 1959
- [Background] Rāzī ABM ibn Z, Arberry AJ. The Spiritual Physick of Rhazes. Butler & Tanner Ltd.; 1950.